CLINICAL TRIAL: NCT06572904
Title: Effect of Intraarticular Injection of Tenoxicam and Hyaluronic Acid Versus Platelet-Rich Plasma and Hyaluronic Acid in Temporomandibular Joint Internal Derangement
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TMJ ID
Record Dates: First submitted 2024-08-23; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Temporomandibular Joint Internal Derangement
Keywords: Tenoxicam; ID; PRP; TMD
MeSH Terms: interventions — Hyaluronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- patients will receive a mixture of tenoxicam and HA. (Experimental): The injection point will be marked Patients will be instructed to open their mouths widely and maintain the mandible in a protruded position A mixture of 1mm of TX and 1ml of HA will be slowly injected intra-articular at the point of entry.
  Interventions: Drug: Tenoxicam Injectable Product; Drug: Hyaluronic Acid 20 MG/1 ML Injection Gel/Jelly
- patients will receive a mixture of PRP and HA. (Experimental): 10 ml of the patient's blood from the ulnar vein into a sterile glass tube containing sodium citrate as an anticoagulant. After mixing the blood with the citrate, using rotating movements, the tubes will be centrifuged at 1500 rpm for 6 min.The injection point will be marked Patients will be instructed to open their mouths widely and maintain the mandible in a protruded position mixture of 1-ml of PRP and 1-ml of HA will be slowly injected intra-articular at the point of entry.
  Interventions: Drug: Hyaluronic Acid 20 MG/1 ML Injection Gel/Jelly

INTERVENTIONS:
Drug: Tenoxicam Injectable Product — (EPICOTIL® Tenoxicam 20 mg , Manufactured by: EGYPTIAN INTERNATIONAL PHARMACEUTICAL INDUSTRIES COMPANY, ReStore at a temperature not exceeding 30°C.)
  Arms: patients will receive a mixture of tenoxicam and HA.
Drug: Hyaluronic Acid 20 MG/1 ML Injection Gel/Jelly — * (Hyalubrix® hyaluronic acid sodium salt 30 MG/2 ML, manufactured by Fidia SPA,Italy, stored at temperature > 25 °C)

SUMMARY:
To compare the effect of intraarticular injection of Tenoxicam and Hyaluronic acid Versus Platelet-rich plasma and Hyaluronic acid in the management of patients with TMJ internal derangement with reduction.

DETAILED DESCRIPTION:
The temporomandibular joint (TMJ) is a bilateral synovial joint located on both sides of the craniomandibular complex, which is involved in chewing, swallowing, speech, and other automatic movements such as yawning, grinding, or clenching; therefore, resting the joint is challenging under normal physiological conditions, except for clamping.Consequently, TMJ pathophysiology significantly impacts individuals' ability to perform basic daily life activities and vital functions.

Temporomandibular disorders (TMDs) are characterized by several symptoms, such as pain or tiredness in the muscles of the face, soreness in the orofacial region, tenderness in the muscles, restricted jaw motion, noise at the joint, hindered jaw function, alteration or diversion, rigidity, soreness, and locking brought on by muscle spasm. TMD may also be accompanied by other neurological symptoms such as headaches, vertigo, heaviness, and impaired vision.

Pain, clicking, a misaligned jaw, and restricted jaw movement are typical symptoms of TMJ ID. The incidence of TMJ pain is shown to affect 9-15% of women and 3-10% of males in the adult population, The disease more frequently affects young persons as opposed to the degenerative lesions of the major joints, This makes TMD a significant social issue that has an impact on people's quality of life.

The primary goal of TMJID treatment is to alleviate pain, restore mandibular functions (mastication and speech), and enhance quality of life.Different therapies, including conservative treatment, minimally invasive surgical operations, and invasive surgical operations, have been widely tested to treat TMD.

Various non-surgical approaches, such as reassurance, physiotherapy, pharmacotherapy, and occlusal splint treatment, have been used to treat TMJID. Minimally invasive treatment approaches for TMJID- include arthrocentesis and intra-articular injections.

Tenoxicam (TX) is a NSAID that is used systemically or locally in joint diseases such as acute or chronic inflammatory rheumatoid arthritis and osteoarthritis.It has been reported that its long-lasting analgesic and anti-inflammatory effects are higher in intra-articular administration than in oral and intravenous administrations. However, there are few studies on intra-articular injection of tenoxicam in patients with temporomandibular joint disc displacements.

Hyaluronic acid (HA) is a high molecular-weight (high-MW) glycosaminoglycan natural synovial fluid and shares in joint lubrication.HA injections have been widely used in the management of TMJDs, and several studies showed promising results in the improvement of maximum inter-incisal opening (MIO) and pain reduction.

The viscosupplementation concept describes the physical mechanism of action mostly carried out by high-MW HAs and by- products. It is based on modifications to HA molecules to promote elasto-viscosity. While the viscoinduction effect of low MW HA, which results in therapeutic benefits after intra-articular Injection, illustrates the underlying process. As a result, the HA-based formulations recommended for the intra-articular treatment of TMJD may differ from one another.

Platelet-rich plasma (PRP) popularly considered as PRP is a concentration of platelets and related growth factors that may have therapeutic effects by attracting, promoting, and differentiating cells as well as remodeling tissue.PRP increases chondrogenic proliferation and the production of matrix molecules, which facilitates joint movement and preserves the chondral surface's overall structure.

HA and PRP mixture were used in many studies treating TMJ or other joints osteoarthritis, PRP restores intra-articular HA, increases glycosaminoglycan chondrocyte synthesis, balances joint angiogenesis, and provides a scaffold for stem cell migration.

To the best of our knowledge, no study up to date has compared the effect of intra-articular injection of a mixture of Tenoxicam and Hyaluronic acid. So, the purpose of this study will be to compare the effect of intra- articular injection of a mixture of (TX and HA) versus (PRP and HA) in the management of patients with TMJ internal derangement with reduction.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age must be (18 -45).
2. Patients have painful joint, clicking sound, with or without limited mouth opening.
3. patients are unresponsive to conservative treatment.
4. Patient's ability and desire to complete the treatment protocol and follow-up visits.
5. Patients with internal derangement with reduction confirmed by MRI imaging.

Exclusion Criteria:

1. Patient with an inflammatory or connective tissue disease
2. Patient with previous invasive TMJ surgical procedure.
3. Neurologic disorders
4. History of injection of any substance into the target TMJ during previous 6 months.
5. History of drug allergy.
6. Patient with a history of bony or fibrous adhesion.
7. Malignant disease in the head and neck region.
8. TMJ Internal derangement without reduction.
9. Patients respond to conservative treatment. 10.Patient with a psychological problem

11.Patients having gross mechanical restrictions and condylar fracture

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2024-10-20 (Estimated); Study Completion 2024-11-20 (Estimated)

PRIMARY OUTCOMES:
Intracapsular Pain and pain during movement | at 1 week, 4, 12, and 24 weeks
  Pain intensity will be measured by VAS score. Zero score for no pain and 10 score for worst pain experienced
Clicking sound | at 1 week, 4, 12, and 24 weeks
  Clicking sound will be assessed as to its presence = 1 or absence =0.
Maximum inter-incisal opening (MIO) | at 1 week, 4, 12, and 24 weeks
  Maximum inter-incisal opening (MIO): was measured by Vernier caliper as the vertical distance in millimeters between the maxillary and mandibular incisal edges of the central incisors.

SECONDARY OUTCOMES:
Magnetic Resonance Imaging (MRI) evaluation | will be done at 24 weeks postoperatively
  Magnetic resonance imaging (MRI) (open and closed) will be done for all patients to diagnose the patients with internal derangement with reduction The MRI protocol included bilateral sagittal oblique proton-density images of the right and left sides in both the closed-mouth (maximum intercuspation) and maximum mouth opening positions.

CONTACTS AND LOCATIONS:
Overall Officials: Sally Awad, Prof, Principal Investigator — Professor of Oral and Maxillofacial Surgery Faculty of Dentistry - Mansoura University; Amira Attia, Dr, Study Director — Lecturer of Oral and Maxillofacial Surgery Faculty of Dentistry- Mansoura University; Manar Mansour, Dr, Study Director — Lecturer of Diagnostic and Interventional Radiology Faculty of Medicine- Mansoura University
Locations (1):
- Mansoura university, Al Mansurah, Egypt

REFERENCES:
- [Background] Lomas J, Gurgenci T, Jackson C, Campbell D. Temporomandibular dysfunction. Aust J Gen Pract. 2018 Apr;47(4):212-215. doi: 10.31128/AFP-10-17-4375. PMID 29621862
- [Background] Ingawale S, Goswami T. Temporomandibular joint: disorders, treatments, and biomechanics. Ann Biomed Eng. 2009 May;37(5):976-96. doi: 10.1007/s10439-009-9659-4. Epub 2009 Feb 28. PMID 19252985
- [Background] Gencer ZK, Ozkiris M, Okur A, Korkmaz M, Saydam L. A comparative study on the impact of intra-articular injections of hyaluronic acid, tenoxicam and betametazon on the relief of temporomandibular joint disorder complaints. J Craniomaxillofac Surg. 2014 Oct;42(7):1117-21. doi: 10.1016/j.jcms.2014.01.041. Epub 2014 Feb 4. PMID 24853591
- [Background] Al-Delayme RMA, Alnuamy SH, Hamid FT, Azzamily TJ, Ismaeel SA, Sammir R, Hadeel M, Nabeel J, Shwan R, Alfalahi SJ, Yasin A. The Efficacy of Platelets Rich Plasma Injection in the Superior Joint Space of the Tempromandibular Joint Guided by Ultra Sound in Patients with Non-reducing Disk Displacement. J Maxillofac Oral Surg. 2017 Mar;16(1):43-47. doi: 10.1007/s12663-016-0911-9. Epub 2016 Jun 10. PMID 28286383
- [Background] Nitzan DW, Dolwick MF, Martinez GA. Temporomandibular joint arthrocentesis: a simplified treatment for severe, limited mouth opening. J Oral Maxillofac Surg. 1991 Nov;49(11):1163-7; discussion 1168-70. doi: 10.1016/0278-2391(91)90409-f. PMID 1941330
- [Background] Israel HA. Internal Derangement of the Temporomandibular Joint: New Perspectives on an Old Problem. Oral Maxillofac Surg Clin North Am. 2016 Aug;28(3):313-33. doi: 10.1016/j.coms.2016.03.009. PMID 27475509
- [Background] Xu J, Ren H, Zhao S, Li Q, Li C, Bao G, Kang H. Comparative effectiveness of hyaluronic acid, platelet-rich plasma, and platelet-rich fibrin in treating temporomandibular disorders: a systematic review and network meta-analysis. Head Face Med. 2023 Aug 26;19(1):39. doi: 10.1186/s13005-023-00369-y. PMID 37633896
- [Background] Sousa BM, Lopez-Valverde N, Lopez-Valverde A, Caramelo F, Fraile JF, Payo JH, Rodrigues MJ. Different Treatments in Patients with Temporomandibular Joint Disorders: A Comparative Randomized Study. Medicina (Kaunas). 2020 Mar 5;56(3):113. doi: 10.3390/medicina56030113. PMID 32151101
- [Background] Attia AAMM, Awad SS. Hyaluronic Acid and Platelet-Rich Plasma Mixture Versus Hyaluronic Acid and Corticosteroid in the Treatment of Temporomandibular Joint Internal Derangement: A Comparative Randomized Study. J Maxillofac Oral Surg. 2023 Apr 5;23(2):1-7. doi: 10.1007/s12663-023-01907-6. Online ahead of print. PMID 37362881
- [Background] Mountziaris PM, Kramer PR, Mikos AG. Emerging intra-articular drug delivery systems for the temporomandibular joint. Methods. 2009 Feb;47(2):134-40. doi: 10.1016/j.ymeth.2008.09.001. Epub 2008 Oct 1. PMID 18835358
- [Background] Hosgor H. Is arthrocentesis plus hyaluronic acid superior to arthrocentesis alone in the treatment of disc displacement without reduction in patients with bruxism? J Craniomaxillofac Surg. 2020 Nov;48(11):1023-1027. doi: 10.1016/j.jcms.2020.07.008. Epub 2020 Jul 25. PMID 33028488
- [Background] Danieli MV, Cavazzani Neto A, Herrera PA. Intra-articular bupivacaine or bupivacaine and morphine after ACL reconstruction. Acta Ortop Bras. 2012;20(5):258-61. doi: 10.1590/S1413-78522012000500002. PMID 24453613
- [Background] Talu GK, Ozyalcin S, Koltka K, Erturk E, Akinci O, Asik M, Pembeci K. Comparison of efficacy of intraarticular application of tenoxicam, bupivacaine and tenoxicam: bupivacaine combination in arthroscopic knee surgery. Knee Surg Sports Traumatol Arthrosc. 2002 Nov;10(6):355-60. doi: 10.1007/s00167-002-0306-y. Epub 2002 Aug 7. PMID 12444514
- [Background] Bayramoglu Z, Yavuz GY, Keskinruzgar A, Koparal M, Kaya GS. Does intra-articular injection of tenoxicam after arthrocentesis heal outcomes of temporomandibular joint osteoarthritis? A randomized clinical trial. BMC Oral Health. 2023 Mar 8;23(1):131. doi: 10.1186/s12903-023-02852-z. PMID 36890529
- [Background] Gigante A, Callegari L. The role of intra-articular hyaluronan (Sinovial) in the treatment of osteoarthritis. Rheumatol Int. 2011 Apr;31(4):427-44. doi: 10.1007/s00296-010-1660-6. Epub 2010 Nov 28. PMID 21113807
- [Background] Ghosh P, Guidolin D. Potential mechanism of action of intra-articular hyaluronan therapy in osteoarthritis: are the effects molecular weight dependent? Semin Arthritis Rheum. 2002 Aug;32(1):10-37. doi: 10.1053/sarh.2002.33720. PMID 12219318
- [Background] Marx RE. Platelet-rich plasma: evidence to support its use. J Oral Maxillofac Surg. 2004 Apr;62(4):489-96. doi: 10.1016/j.joms.2003.12.003. No abstract available. PMID 15085519
- [Background] Abrams GD, Frank RM, Fortier LA, Cole BJ. Platelet-rich plasma for articular cartilage repair. Sports Med Arthrosc Rev. 2013 Dec;21(4):213-9. doi: 10.1097/JSA.0b013e3182999740. PMID 24212369
- [Background] Samiee A, Sabzerou D, Edalatpajouh F, Clark GT, Ram S. Temporomandibular joint injection with corticosteroid and local anesthetic for limited mouth opening. J Oral Sci. 2011 Sep;53(3):321-5. doi: 10.2334/josnusd.53.321. PMID 21959659
- [Background] Spakova T, Rosocha J, Lacko M, Harvanova D, Gharaibeh A. Treatment of knee joint osteoarthritis with autologous platelet-rich plasma in comparison with hyaluronic acid. Am J Phys Med Rehabil. 2012 May;91(5):411-7. doi: 10.1097/PHM.0b013e3182aab72. PMID 22513879